CLINICAL TRIAL: NCT07076901
Title: Effectiveness of Prehabilitation Strategies in Enhancing Recovery and Postoperative Outcomes in Laparoscopic Sleeve Gastrectomy Patients
Brief Title: Prehabilitation Strategies for Patients Undergoing Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yankai Zhao, Principal Investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023S00457
Record Dates: First submitted 2025-07-02; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Obesity &Amp; Overweight
Keywords: Prehabilitation strategy; laparoscopic sleeve gastrectomy; weight loss outcomes; quality of life; postoperative complications
MeSH Terms: conditions — Obesity; Overweight; Postoperative Complications | interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation Group (Prehabilitation) (Experimental): Participants received a multi-component prehabilitation program for 5-7 days before surgery. The program consisted of structured psychological, exercise, and lifestyle interventions administered by a multidisciplinary team, in addition to routine perioperative care.
  Interventions: Behavioral: Psychological Support; Behavioral: Supervised Exercise Program; Behavioral: Lifestyle and Dietary Modification
- Control Group (Routine Care) (Active Comparator): Participants received standard hospital perioperative care as per institutional protocol, without the specific, structured prehabilitation interventions provided to the observation group.
  Interventions: Other: Routine Perioperative Care

INTERVENTIONS:
Behavioral: Psychological Support — A structured psychological intervention aimed at alleviating preoperative anxiety. It included one-on-one counseling, providing detailed information about the surgical procedure, introducing relaxation techniques and music therapy, and sharing success stories from previous patients to boost confidence. Support was provided via phone or WeChat video by a qualified psychological counselor.
  Arms: Observation Group (Prehabilitation)
Behavioral: Supervised Exercise Program — A daily guided exercise regimen including two components: 1) General physical conditioning consisting of at least 40 minutes of moderate-intensity aerobic and resistance training (e.g., brisk walking, jogging, cycling). 2) Respiratory function training consisting of abdominal breathing (5 times/hour) and balloon-blowing exercises (10 times/day). Patient adherence was monitored daily via a WeChat group.
  Arms: Observation Group (Prehabilitation)
Behavioral: Lifestyle and Dietary Modification — Focused on optimizing preoperative habits. Nutritional guidance involved a high-protein, high-vitamin diet with six smaller, frequent meals per day to adapt to post-surgery conditions. Lifestyle guidance included advising smoking and alcohol cessation and ensuring 6-8 hours of sleep per night. Daily dietary and sleep status were reported and monitored via a WeChat group.
  Arms: Observation Group (Prehabilitation)
Other: Routine Perioperative Care — Consisted of standard care practices before, during, and after surgery. Preoperative care included health education and fasting instructions. Intraoperative care included body temperature maintenance and vital signs monitoring. Postoperative care included 12-hour ECG monitoring, gradual reintroduction of a clear liquid diet 24 hours post-surgery, encouragement of early mobilization, and standard nursing for catheters and wounds.
  Arms: Control Group (Routine Care)

SUMMARY:
This study aims to evaluate the effectiveness of prehabilitation strategies in patients undergoing laparoscopic sleeve gastrectomy (LSG). The study compares a group receiving prehabilitation (including exercise, nutritional, and psychological support) with a control group receiving routine care. The primary goal is to determine if prehabilitation improves postoperative recovery, enhances weight loss, improves quality of life, and reduces complications.

DETAILED DESCRIPTION:
Obesity is a significant global health issue, and laparoscopic sleeve gastrectomy (LSG) is a common surgical treatment. However, the procedure is invasive and can cause physical and psychological stress, impacting postoperative recovery. Prehabilitation, a process of enhancing a patient's functional capacity before surgery, has shown promise in various surgical fields. This study investigates a "triad prehabilitation management mode," incorporating psychological intervention, nutritional support, and exercise training for patients undergoing LSG. This prospective, randomized controlled trial enrolled 120 patients assigned to either a prehabilitation group or a control group. The prehabilitation group received a structured program of exercise, nutritional guidance, and psychological support for 5-7 days before surgery, in addition to routine care. The control group received routine care only. The study hypothesizes that the prehabilitation strategy will lead to faster gastrointestinal function recovery, better weight loss outcomes, improved quality of life, and a lower rate of postoperative complications compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* Obesity, defined by a body mass index (BMI) ≥35 kg/m².
* Age between 18 and 50 years.
* Failure of non-surgical weight loss methods.
* Surgical eligibility for LSG based on clinical assessment.
* Willingness to participate in the study and sign an informed consent form.

Exclusion Criteria:

* Incomplete clinical data.
* Inability to strictly adhere to dietary instructions.
* Inability to complete follow-up visits.
* Secondary obesity.
* Presence of mental disorders, cognitive impairment, or consciousness disturbance.
* Planned pregnancy within 1 year post-surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Time to recovery of bowel motility | Perioperative
  Time in days from surgery until the first audible bowel sounds.
Time to first flatus | Perioperative
  Time in hours/days from surgery until the patient's first passage of flatus.
Time to first bowel movement | Perioperative
  Time in days from surgery until the patient's first bowel movement.
Time to first eating | Perioperative
  Time in hours/days from surgery until the patient starts clear liquids.
Duration of hospital stay | Perioperative
  Total length of stay in the hospital, measured in days.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and 6 months post-surgery
  Change in BMI (kg/m²) from baseline to 6 months post-surgery.
Change in Waist Circumference | Baseline and 6 months post-surgery
  Change in waist circumference (cm) from baseline to 6 months post-surgery.
Quality of Life Score | Baseline and 6 months post-surgery
  Change in score on the Medical Outcomes Study Short Form 36 (MOS SF-36) Health Survey. The scale assesses eight dimensions, with higher scores indicating better quality of life.
Incidence of Postoperative Complications | Perioperative and 6 months post-surgery
  The percentage of patients experiencing complications such as abdominal distention, bleeding, and anastomotic leak.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China